CLINICAL TRIAL: NCT04420767
Title: The Effect of Brain Neuromodulation on Food Cravings, Cognitive Control and Food Addiction Scales in Overweight/Obese Women Using tDCS
Brief Title: The Effect of Brain Stimulation (tDCS) in Food Cravings Control in Overweight/Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Claudia P. Sanmiguel, MD, Health Sciences Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#15-001929
Record Dates: First submitted 2017-04-21; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Obesity
Keywords: food cravings; neuromodulation; brain; cognitive control; tDCS; prefrontal cortex; MRI; food addiction
MeSH Terms: conditions — Obesity; Food Addiction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS and Go-No Go task (Experimental): Certain randomly assigned participants will receive tDCS to the DLPFC for 8 daily 20-minute sessions, with a TDCS amplitude of 2 mAmps.
  During the tDCS session, individuals will perform a 10-min computerized Go-No Go task
  Interventions: Device: tDCS; Behavioral: Go-No GO task
- Sham brain stimulation and Go-No Go task (Sham Comparator): Certain randomly assigned participants will receive Sham Stimulation to the DLPFC for 8 daily 20-min sessions. The Sham stimulation is an inactive form of stimulation.
  During the sham brain stimulation session, individuals will perform a 10-min computerized Go-No Go task
  Interventions: Device: Sham brain stimulation; Behavioral: Go-No GO task

INTERVENTIONS:
Device: tDCS — Individuals undergo 20min daily sessions receiving actual tDCS to the brain (to the right DLPFC: dorsolateral prefrontal cortex)
  Other Names: Real brain stimulation
  Arms: tDCS and Go-No Go task
Device: Sham brain stimulation — Individuals undergo 20min daily sessions receiving sham stimulation to the brain (to the right DLPFC: dorsolateral prefrontal cortex)
  Arms: Sham brain stimulation and Go-No Go task
Behavioral: Go-No GO task — During the brain stimulation sessions, all individuals will be asked to perform a 10 min-computerized task related to inhibitory control (Go-No Go)

SUMMARY:
This study is a randomized clinical trial to test the effect of a type of non-invasive brain stimulation on the response to a behavioral intervention designed to enhance cognitive control over food cravings in obese and overweight women. The brain stimulation is called transcranial Direct Current Stimulation (tDCS). All eligible participants will engage in a behavioral intervention known to enhance control over food cravings and will be randomly assigned to receive either tDCS or sham stimulation to the prefrontal cortex of the brain.

DETAILED DESCRIPTION:
This study is a randomized clinical trial to test the effect of a type of non-invasive brain stimulation on the response to a behavioral intervention designed to enhance cognitive control over food cravings in obese and overweight women. The brain stimulation is called transcranial Direct Current Stimulation (tDCS) which is a form of stimulation that delivers a low amplitude electrical current to the brain via the scalp (i.e. trans-cranial) to modify brain activity.

All eligible participants will engage in a behavioral intervention (Go-No Go task), known to enhance control over food cravings, and will be randomly assigned to receive either tDCS or sham stimulation to the right prefrontal cortex of the brain during 8 20-min daily sessions.

Primary outcome: score changes in eating behaviors scales (YFAS and TFEQ), scales will be applied at baseline and at the end of the 8 brain stimulation sessions.

Secondary outcomes: changes in diet, brain function (brain MRI/MRS) Other outcomes: food cravings scales and impulse control scales and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

BMI between 28 and 40 kg/m2 high scores in the Yale-Food Addiction-Scale right-handed

Exclusion Criteria:

* History of anorexia nervosa or bulimia or binge eating disorder
* Any contraindication to undergo MRI
* Use of psychotropic medications and/or opiate pain medications.
* Current or past alcohol or drug abuse problem or smoking
* Pregnancy
* Current use of weight loss medication or currently participating in a weight loss program.
* History of seizures, epilepsy or factors/medications associated with lowered seizure threshold.
* History of brain disease or major neurological disorder or mental disorder
* History of brain surgery or history of loss of consciousness >15 min
* History of major gastrointestinal surgery including weight loss surgery
* History of endocrine imbalances including diabetes, thyroid disease, Cushing's disease, metabolic syndrome and polycystic ovary.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Yale Food Addiction Scale scores | Scores measured at baseline and at up-to 2 weeks after the intervention
  Yale Food Addiction Scale (YFAS26) that is a 25-item measure developed to measure food addiction. Score range: 0 to 7. Higher scores in the scale mean more symptoms resembling food addiction (worse).
Change in Three-Factor Eating Questionnaire scores | Scores measured at baseline and at up-to 2 weeks after the intervention
  Three-Factor Eating Questionnaire is a validated scale that is designed to measure 3 dimensions of human eating behavior: cognitive restraint of eating (Factor I), disinhibition (Factor II), and hunger (Factor III). The minimum score for factors I-II-III is therefore 0-0-0, and maximum possible score is 20-16-15. Higher scores in the respective scales are indicative of greater cognitive restraint (better), uncontrolled (worse), or emotional eating (worse).

SECONDARY OUTCOMES:
Change in brain neural activity by functional Magnetic Resonance Imaging ( fMRI) | Brain function at baseline and up-to 2 weeks after the intervention
  Significant change in brain activity of the prefrontal cortex (area involved in the inhibitory control of food intake) measured by modification of BOLD (Blood-Oxygen-Level-Dependent) signal in fMRI evoked responses to visual food-cues
Change in Brain metabolites concentrations by Magnetic Resonance Spectroscopy (MRS) | Brain MRS at baseline and up-to 2 weeks after the intervention
  Significant change in brain metabolites concentration at the prefrontal cortex (area involved in the inhibitory control of food intake) measured with Magnetic Resonance spectroscopy

OTHER OUTCOMES:
Diet (3-day food intake record) | Values measured at baseline and at up-to 2 weeks after the intervention
  3-day food intake record: individuals will record everything they eat and drink for 3 days. To assess calorie intake and macro nutrients
Change in Yale Food Addiction Scale scores at 3-months post-intervention | At 3-months after intervention
  Yale Food Addiction Scale (YFAS26) that is a 25-item measure developed to measure food addiction. Score range: 0 to 7. Higher scores in the scale mean more symptoms resembling food addiction (worse).
Change in Three-Factor Eating Questionnaire scores at 3-months post-intervention | At 3-months after intervention
  Three-Factor Eating Questionnaire is a validated scale that is designed to measure 3 dimensions of human eating behavior: cognitive restraint of eating (Factor I), disinhibition (Factor II), and hunger (Factor III). The minimum score for factors I-II-III is therefore 0-0-0, and maximum possible score is 20-16-15. Higher scores in the respective scales are indicative of greater cognitive restraint (better), uncontrolled (worse), or emotional eating (worse).
Cognitive function assessment | Measured at baseline and up-to 2 weeks after the intervention
  Multiple Abilities Self-Report Questionnaire (MASQ), a self-report measure comprising items from five cognitive domains; language, visuo-perceptual, verbal memory, visual memory, and attention. The maximum score for the whole scale is 190 points. Higher scores correlate with better function.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia P Sanmiguel, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States